CLINICAL TRIAL: NCT04456296
Title: An Open-Label, Randomized, Parallel-Group, Three Treatment Arm, Multicenter Study on Hypogonadal Males to Evaluate the Effect on 24-Hour Ambulatory Blood Pressure After 16-Week Continuous Treatment With Marketed Testosterone Products
Brief Title: A Study of the Effect of Testosterone Replacement Therapy on Blood Pressure in Adult Male Participants With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3000-101
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hypogonadism; Hypogonadism, Male; Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism; Eunuchism | interventions — testosterone undecanoate; Testosterone Propionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AVEED (Testosterone Undecanoate Injection) (Active Comparator): Fixed dosage level of 750 milligrams (mg)/3 milliliters (mL) administered by intramuscular injections.
  Interventions: Drug: Aveed Injectable Product
- FORTESTA (Testosterone Gel) (Active Comparator): 40 mg once daily topical gel administration.
  Interventions: Drug: Fortesta
- TESTIM (Testosterone Gel) (Active Comparator): 50 mg once daily topical gel administration.
  Interventions: Drug: Testim

INTERVENTIONS:
Drug: Aveed Injectable Product — Testosterone undecanoate administered by intramuscular injections.
  Other Names: Testosterone undecanoate
  Arms: AVEED (Testosterone Undecanoate Injection)
Drug: Fortesta — Testosterone gel administered topically. The daily dose of the study drug will be titrated for each participant, according to approved dosage and administration instructions, until the circulating testosterone concentrations of the participant reaches normal concentrations (300-1000 ng/dL).
  Other Names: Testosterone gel
  Arms: FORTESTA (Testosterone Gel)
Drug: Testim — Testosterone gel administered topically. The daily dose of the study drug will be titrated for each participant, according to approved dosage and administration instructions, until the circulating testosterone concentrations of the participant reaches normal concentrations (300-1000 ng/dL).
  Other Names: Testosterone gel
  Arms: TESTIM (Testosterone Gel)

SUMMARY:
Testosterone is the principal androgen produced by the male testes. Male Hypogonadism is the result of inadequate production of testosterone by the Leydig cells of the testes and is reflected by total serum concentrations of testosterone of < 300 nanograms (ng)/deciliters (dL), with no discernible diurnal pattern. The etiology of hypogonadism may be primary or secondary. The treatment of males with primary, and in some cases, secondary hypogonadism includes administration of testosterone.

Testim® and Fortesta® are topical gels that when applied daily help to increase the total testosterone levels in the blood through skin absorption. Aveed® is an injectable form of testosterone treatment and participants randomized to this treatment arm will receive 3 injections over the course of 16 weeks.

This study is designed to evaluate the effect on blood pressure of approved testosterone products (Testim®, Fortesta®, and Aveed®) after 16 weeks of therapy using 24-hour ambulatory blood pressure to reveal shifts in blood pressure levels.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of primary hypogonadism or hypogonadotropic hypogonadism.
2. Have a total serum testosterone at screening < 300 ng/dL based on 2 blood samples obtained at 10 am (+/-2 hours) on 2 separate occasions at least 48 hours apart
3. Be naïve to androgen replacement or washout of 12 weeks following intramuscular androgen injections; 4 weeks following topical or buccal, nasal, or oral androgens.
4. Have a screening blood pressure at rest of less than 140 millimeters of mercury (mm Hg) for systolic blood pressure and less than 90 mm Hg for diastolic blood pressure.
5. Be judged to be in good health.
6. Participants enrolled in the Testim or Fortesta treatment arms: participants agree to take necessary precautions to avoid skin-to-skin contact and potential transfer and if male use effective contraception.
7. Be willing and able to cooperate with the requirements of the study.

Exclusion Criteria:

1. Is from a vulnerable population, as defined by the US Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board/Independent Ethics Committee (IRB/IEC).
2. Has a history of significant sensitivity or allergy to the study drugs, including androgens, or product excipients.
3. Has a history of or medical examination findings renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric conditions, cardiovascular disease/dysrhythmia) or any other condition(s) that restricts study participation.
4. Has clinically significant changes in any medications (including dosages) or medical conditions in the 28 days prior to screening
5. Is not on a stable medication regimen for at least 3 months for the treatment of a chronic condition.
6. Has had a cardiovascular and/or cerebrovascular event within the last 6 months.
7. Needs blood pressure cuff size larger than 50 centimeters.
8. Works a night shift or performs heavy manual labor.
9. Has any known contraindication(s) to active study treatment including, but not limited to: known or suspected carcinoma of the prostate or breast, previous history of cancer (except basal cell carcinoma of the skin) liver disease, active deep vein thrombosis, atrial fibrillation, untreated sleep apnea, or is immune compromised.
10. Uses known inhibitors (for example, ketoconazole) or inducers of cytochrome P450 3A (for example, dexamethasone, phenytoin, rifampin, carbamazepine) of cytochrome P450 3A (CYP3A) within 30 days prior to study drug administration and through the end of the study.

    1. Uses any of the above listed drugs within 5 half lives of the last dose in the past 6 months prior to study drug administration.
    2. Has received any of the above listed drugs by injection within 30 days or 10 half lives (whichever is longer) prior to study drug administration.
    3. Uses nutraceuticals or homeopathic compounds which have a known effect on blood pressure.
11. Has a history of drug or alcohol abuse within 6 months prior to study drug administration.
12. Has untreated moderate to severe depression.
13. Has any skin lesions/cuts/injury at the application site that prohibits topical application and/or intramuscular injection of study drug.
14. Has suspected reversible hypogonadism.
15. Donated blood or blood products or experienced significant blood loss within 90 days prior to study drug administration.
16. Intends to conceive at any time during the study.
17. Donated bone marrow within 6 months prior to study drug administration.
18. Has participated in a previous investigational study or received treatment with an investigational product within 30 days of screening.
19. Has a diagnosis of, is undergoing therapy for, or has received therapy for a hematologic malignancy in the 5 years prior to screening.
20. Has a history of substance abuse or is taking any substance of abuse (Note: participants on a stable dose of any medications that have been prescribed by a healthcare practitioner for a properly documented medical condition are exempt).
21. Abnormal electrocardiogram (ECG) (QT prolongation with QTc ≥450 milliseconds).
22. Has evidence of abnormalities on physical examination, vital signs, ECG, or clinical lab values, unless judged to be clinically insignificant by the investigator
23. Has any other condition that, in the investigator's opinion, might indicate the participant to be unsuitable for the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 673 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hernandez, Study Director — Endo Pharmaceuticals
Locations (35):
- United States (35):
  - Endo Clinical Trial Site #8, Birmingham, Alabama
  - Endo Clinical Trial Site #22, Tucson, Arizona
  - Endo Clinical Trial Site #15, North Little Rock, Arkansas
  - Endo Clinical Trial Site #32, Bell Gardens, California
  - Endo Clinical Trial Site #33, Canoga Park, California
  - Endo Clinical Trial Site #30, Beverly Hills, Florida
  - Endo Clinical Trial Site #12, Boynton Beach, Florida
  - Endo Clinical Trial Site #34, Boynton Beach, Florida
  - Endo Clinical Trial Site #29, Fleming Island, Florida
  - Endo Clinical Trial Site #26, Miami, Florida
  - Endo Clinical Trial Site #2, Miami, Florida
  - Endo Clinical Trial Site #28, Miami, Florida
  - Endo Clinical Trial Site #10, Miami Beach, Florida
  - Endo Clinical Trial Site #18, Miami Gardens, Florida
  - Endo Clinical Trial Site #3, Oviedo, Florida
  - Endo Clinical Trial Site #4, Pembroke Pines, Florida
  - Endo Clinical Trial Site #11, Pompano Beach, Florida
  - Endo Clinical Trial Site #23, West Palm Beach, Florida
  - Endo Clinical Trial Site #16, Chicago, Illinois
  - Endo Clinical Trial Site #27, Glen Burnie, Maryland
  - Endo Clinical Trial Site #17, Towson, Maryland
  - Endo Clinical Trial Site #35, East Orange, New Jersey
  - Endo Clinical Trial Site #9, Garden City, New York
  - Endo Clinical Trial Site #7, New York, New York
  - Endo Clinical Trial Site #25, Winston-Salem, North Carolina
  - Endo Clinical Trial Site #5, Dayton, Ohio
  - Endo Clinical Trial Site #13, Bala-Cynwyd, Pennsylvania
  - Endo Clinical Trial Site #19, Houston, Texas
  - Endo Clinical Trial Site #31, Houston, Texas
  - Endo Clinical Trial Site #20, Houston, Texas
  - Endo Clinical Trial Site #21, Missouri City, Texas
  - Endo Clinical Trial Site #1, San Antonio, Texas
  - Endo Clinical Trial Site #14, Rutland, Vermont
  - Endo Clinical Trial Site #6, Charlottesville, Virginia
  - Endo Clinical Trial Site #24, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- AVEED® (Testosterone Undecanoate Injection): Participants received 750 milligrams (mg)/3 milliliters (mL) of injection administered by intramuscular route on Days 2, 30 and 100.
- FORTESTA® (Testosterone Gel): Participants received 40 mg once daily topical gel application starting from Day 2. Participants were followed up on Day 16, Day 37, Day 67, and Day 97.
- TESTIM® (Testosterone Gel): Participants received 50 mg once daily topical gel application starting from Day 2. Participants were followed up on Day 16, Day 37, Day 67, and Day 97.
Period: Overall Study
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Started | 224 | 224 | 225
Safety Population (All participants who received at least 1 dose of study drug.) | 222 | 223 | 225
Intent-to-Treat (ITT) Population (All randomized participants who had at least 1 dose of study drug.) | 222 | 223 | 225
Full Analysis Set (All randomized participants who had at least 1 dose/injection of study medication and valid Baseline and end of study Ambulatory Blood Pressure Monitoring (ABPM) assessments.) | 140 | 133 | 134
Completed | 202 | 194 | 192
Not Completed | 22 | 30 | 33
Not completed — Withdrawal by Subject | 14 | 21 | 21
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 5 | 6
Not completed — Other than specified | 0 | 1 | 4
Not completed — Randomized, not treated | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose/injection of study intervention.
Groups:
- AVEED® (Testosterone Undecanoate Injection): Participants received 750 mg/3 mL of injection administered by intramuscular route on Days 2, 30 and 100.
- Total: Total of all reporting groups
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel) | Total
Number analyzed (Participants) | 222 | 223 | 225 | 670
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (10.10) | 56.3 (10.78) | 58.4 (10.22) | 58.2 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 222 | 223 | 225 | 670
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 92 | 79 | 242
  Not Hispanic or Latino | 151 | 131 | 146 | 428
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 8 | 1 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
  Black or African American | 37 | 41 | 43 | 121
  White | 174 | 179 | 168 | 521
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
24-Hour Average Systolic Ambulatory Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: ITT Population included all randomized participants who received at least 1 dose/injection of study medication.
  mmHg | 124.90 (12.178) | 123.95 (11.499) | 124.45 (12.505) | 124.43 (12.058)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-Hour Average Systolic Ambulatory Blood Pressure to End of Study (EOS)
Description: The mean change from Baseline to EOS in 24-hour average systolic ambulatory blood pressure, for each treatment group was analyzed using an analysis of covariance (ANCOVA) model with treatment and study center (pooled centers) as fixed effects, Baseline 24-hour average systolic ambulatory blood pressure as covariate. EOS for the Aveed arm was Day 107 and EOS for Fortesta and Testim, was Day 114.
Time Frame: Baseline (Day 1), EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
millimeters of mercury (mmHg) | 2.77 [0.95 to 4.59] | 2.78 [0.86 to 4.69] | 2.15 [0.28 to 4.03]

2. Secondary Outcome: Change From Baseline in 24-Hour Average Mean Arterial Pressure (MAP) to EOS
Description: The mean change from Baseline to EOS in 24-hour MAP, for each treatment group was analyzed using an ANCOVA model with treatment and study center (pooled centers) as fixed effects, Baseline 24-hour MAP as covariate.EOS for the Aveed arm was Day 107 and EOS for Fortesta and Testim, was Day 114.
Time Frame: Baseline (Day 1), EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
mmHg | 2.13 [0.89 to 3.37] | 1.78 [0.47 to 3.08] | 1.21 [-0.06 to 2.49]

3. Secondary Outcome: Change From Baseline in 24-Hour Average Diastolic Ambulatory Blood Pressure to EOS
Description: The mean change from Baseline to EOS in 24-hour average diastolic ambulatory blood pressure, for each treatment group was analyzed using an ANCOVA model with treatment and study center (pooled centers) as fixed effects, Baseline 24-hour average diastolic ambulatory blood pressure as covariate. EOS for the Aveed arm was Day 107 and EOS for Fortesta and Testim, was Day 114.
Time Frame: Baseline (Day 1), EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
mmHg | 1.85 [0.79 to 2.91] | 1.22 [0.10 to 2.34] | 0.81 [-0.28 to 1.91]

4. Secondary Outcome: Change From Baseline in 24-Hour Average Heart Rate to EOS
Description: The mean change from Baseline to EOS in 24-hour average heart rate, for each treatment group was analyzed using an ANCOVA model with treatment and study center (pooled centers) as fixed effects, Baseline 24-hour average heart rate as covariate. EOS for the Aveed arm was Day 107 and EOS for Fortesta and Testim, was Day 114.
Time Frame: Baseline (Day 1), EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
beats per minute | 2.89 [1.47 to 4.31] | 1.56 [0.07 to 3.06] | 1.84 [0.37 to 3.31]

5. Secondary Outcome: Change From Baseline in 24-Hour Average Pulse Pressure (PP) to EOS
Description: The mean change from Baseline to EOS in 24-hour average PP for each treatment group was analyzed using an ANCOVA model with treatment and study center (pooled centers) as fixed effects, Baseline 24-hour average PP as covariate. EOS for the Aveed arm was Day 107 and EOS for Fortesta and Testim, was Day 114.
Time Frame: Baseline (Day 1), EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
mmHg | 0.80 [-0.41 to 2.0] | 1.49 [0.22 to 2.75] | 1.40 [0.16 to 2.63]

6. Secondary Outcome: Percentage of Participants Taking New Antihypertensive Medications
Description: A new antihypertensive medication was any antihypertensive medication taken on or after the screening Visit through the EOS visit and not taken prior to the screening visit.
Time Frame: EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Number; unit: Percentage of participants
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
Percentage of participants | 1.4 | 1.5 | 2.2

7. Secondary Outcome: Percentage of Participants With Dose Increase From Baseline in Antihypertensive Medications
Description: as for outcome 6
Time Frame: EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Population: Full analysis set included all ITT participants with valid Baseline and EOS ABPM assessments.
Measure: Number; unit: Percentage of participants
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
Number analyzed (Participants) | 140 | 133 | 134
Percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to EOS Visit: up to Day 107 for the Aveed Arm, and up to Day 114 for Fortesta and Testim Arms
Description: All cause-mortality was based on enrolled participants. SAEs and other non-serious AEs were based on the Safety population that included all participants who received at least 1 dose of study drug. Three participants did not receive at least 1 dose of study drug.
Arm/Group | AVEED® (Testosterone Undecanoate Injection) | FORTESTA® (Testosterone Gel) | TESTIM® (Testosterone Gel)
All-Cause Mortality (participants affected / at risk) | 1/224 | 0/224 | 0/225
Serious Adverse Events (participants affected / at risk) | 3/222 | 1/223 | 2/225
Other Adverse Events (participants affected / at risk) | 8/222 | 9/223 | 13/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVEED® (Testosterone Undecanoate Injection) (N=222) | FORTESTA® (Testosterone Gel) (N=223) | TESTIM® (Testosterone Gel) (N=225)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVEED® (Testosterone Undecanoate Injection) (N=222) | FORTESTA® (Testosterone Gel) (N=223) | TESTIM® (Testosterone Gel) (N=225)
Headache (Nervous system disorders) | 1 | 2 | 3
Blood testosterone increased (Investigations) | 0 | 2 | 3
Hypertension (Vascular disorders) | 7 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2002-02-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT04456296/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT04456296/SAP_001.pdf